CLINICAL TRIAL: NCT02480153
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND STUDY ASSESSING THE EFFICACY AND SAFETY OF PF-06410293 AND ADALIMUMAB IN COMBINATION WITH METHOTREXATE IN SUBJECTS WITH MODERATELY TO SEVERELY ACTIVE RHEUMATOID ARTHRITIS WHO HAVE HAD AN INADEQUATE RESPONSE TO METHOTREXATE
Brief Title: A Study Of PF-06410293 (Adalimumab-Pfizer) And Adalimumab (Humira®) In Combination With Methotrexate In Subjects With Active Rheumatoid Arthritis (REFLECTIONS B538-02).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B5381002; B5381002, REFLECTIONS B538-02; 2014-000352-29 (EudraCT Number); ADALIMUMAB (Other: Alias Study Number)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Phase 3; adalimumab; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PF-06410293; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-06410293 (Experimental)
  Interventions: Biological: PF-06410293
- Adalimumab (Active Comparator)
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: PF-06410293 — PF-06410293 will be administered with a uniform dose regimen, which is SC injection at a dose of 40 mg every other week, throughout the study treatment.
  Other Names: Adalimumab-Pfizer
  Arms: PF-06410293
Biological: Adalimumab — Adalimumab will be administered with a uniform dose regimen, which is SC injection at a dose of 40 mg every other week, throughout the study treatment.
  Other Names: Adalimumab-European Union, Humira®
  Arms: Adalimumab

SUMMARY:
The study will assess the efficacy, safety, and immunogenicity of PF-06410293 and adalimumab in combination with methotrexate in subjects with moderately to severly active rheumatoid arthritis who have had an inadequate response to methotrexate.

In an additional optional portion of the study, during open label Treatment Period 3 (TP3), a subset of subjects used a Prefilled Pen (PFP) to administer up to 3 injections of their study treatment (PF-06410293) at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis based on 2010 ACR/EULAR criteria for at least 4 months.
* At least 6 tender (of 68 assessed) and 6 swollen (of 66 assessed) joints at screening and baseline.
* Hs-CRP equal or greater than 8 mg/L.
* Must have received methotrexate for at least 12 weeks and been on a stable dose for at least 4 weeks prior to the first study dose.

Exclusion Criteria:

* Evidence of untreated or inadequately treated latent or active TB.
* Evidence of uncontrolled, clinically significant diseases, including moderate or severe heart failure (NYHA Class III/IV) or malignancy in the previous 5 years.
* History of infection requiring hospitalization or parenteral antimicrobial therapy within 6 months prior to first dose of study drug.
* May have received no more than 2 doses of one biologic therapy (other than adalimumab or lymphocyte depleting therapy).
* Any second DMARD must be washed out prior to the first study dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (183):
- United States (49):
  - ArthroCare, Arthritis Care & Research P.C., Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Associates, PC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates, PC, Phoenix, Arizona
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Westlake Medical Research, Thousand Oaks, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Desert Valley Medical Group, Victorville, California
  - Javed Rheumatology Associates, Inc, Newark, Delaware
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Robert W. Levin, MD, PA, Clearwater, Florida
  - International Medical Research, Daytona Beach, Florida
  - SIMED Arthritis Center, Gainesville, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research, Gainesville, Florida
  - Rheumatology Associates of Central Florida, P.A., Orlando, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Alastair C. Kennedy, MD, Vero Beach, Florida
  - Indian River Primary Care, Vero Beach, Florida
  - St Luke's Intermountain Research Center, Boise, Idaho
  - St Luke' s Clinic, Meridian, Idaho
  - Physician's Clinic of Iowa, P.C., Cedar Rapids, Iowa
  - Graves-Gilbert Clinic Bowling Green, Bowling Green, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Bronson Internal Medicine and Rheumatology, Battle Creek, Michigan
  - North Mississippi Medical Clinics, Inc. - Clinical Research, Tupelo, Mississippi
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Clinical Research, Inc., Omaha, Nebraska
  - Arthritis, Rheumatic & Back Disease Associates, P.A., Voorhees Township, New Jersey
  - Manhattan Medical Research, New York, New York
  - Buffalo Rheumatology and Medicine PLLC, Orchard Park, New York
  - Physicians East PA, Greenville, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research of Reading, LLC, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Regional Medical Clinic - Rheumatology, Rapid City, South Dakota
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta, M.D., Memphis, Tennessee
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - The Clinical Research Institute of Houston, LLC, Houston, Texas
  - Accurate Clinical Research, League City, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Northwest Diagnostic Clinic, PA, Shenandoah, Texas
  - Center for Arthritis and Rheumatic Diseases, P.C., Chesapeake, Virginia
  - Wenatchee Valley Hospitals & Clinics, Wenatchee, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Australia (3):
  - Paradise Arthritis & Rheumatology Pty Ltd, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - RK Will Pty Ltd, Victoria Park, Western Australia
- EDUMED Educação em Saúde S/S Ltda, Curitiba, Paraná, Brazil
- Bulgaria (4):
  - MHAT Plovdiv AD, Plovdiv
  - University Multiprofile Hospital for Active Treatment (UMHAT) Kaspela EOOD, Plovdiv
  - UMHAT "Sv. Ivan Rilski" EAD, Sofia
  - University Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski" EAD, Sofia
- Fundacion Instituto de Reumatologia Fernando Chalem, Bogotá, Colombia
- Czechia (9):
  - Lekarna Na vrsku, Bruntál
  - Revmatologie Bruntal, s.r.o., Bruntál
  - L.K.N. Arthrocentrum, s.r.o., Hlučín
  - Lekarna Vesalion, Ostrava
  - Benu Lekarna, Pardubice
  - CCBR-SYNARC, a.s., Pardubice
  - Revmatologicky ustav, Prague
  - Lekarna Hradebni s.r.o., Uherské Hradiště
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
- Estonia (2):
  - Innomedica OÜ, Tallinn
  - East Tallinn Central Hospital, Tallinn
- Georgia (10):
  - LTD "Unimed Adjara", Batumi, Adjara
  - Unimedi Kakheti Ltd, Telavi Referral Hospital, Telavi, Kakheti
  - V.Tsitlanadze Scientifically-Practical Rheumatology Center LTD, Tbilisi
  - V.Tsitlanadze Scientifically-Practical Rheumatology Center, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic Helsicore", Tbilisi
  - LTD Cardio-Reanimation Center, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - LTD Altravita, Tbilisi
  - LTD.MediClubGeorgia, Tbilisi
  - JSC Medical Corporation Evex, Tbilisi
- Germany (7):
  - Schlosspark-Klinik, Berlin
  - Gemeinschaftspraxis Dr. von Hinüber/Dr. Demary, Hildesheim
  - Klinikum der Universität München, München
  - Praxiszentrum St. Bonifatius, München
  - Rheumapraxis Dr. Martin Welcker und Kollegen, Planegg
  - Knappschaftsklinikum Saar GmbH, Püttlingen
  - Rheumazentrum Ratingen, Ratingen
- Hungary (3):
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Qualiclinic Kft., Budapest
  - Vital Medical Center Orvosi es Fogorvosi Kozpont, Veszprém
- Japan (12):
  - Anjo Kosei Hospital, Anjo-shi, Aichi-ken
  - Inoue Hospital, Takasaki, Gunma
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Katayama Orthopaedic Rheumatology Clinic, Asahikawa, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Matsubara Mayflower Hospital, Katō, Hyōgo
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Saitama Medical Center, Kawagoe, Saitama
  - Hirose Clinic, Tokorozawa, Saitama
  - Kondo clinic for rheumatism and orthopaedics, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
- Lithuania (3):
  - LSMUL Kauno klinikos, Kaunas
  - Klaipedos universitetine ligonine, Klaipėda
  - Vilniaus universiteto ligonines Santariskiu klinikos, Vilnius
- Mexico (2):
  - Consultorio Medico Privado de Reumatologia, Mexicali, Estado de Baja California
  - Consultorio de Reumatologia, Mexico City
- New Zealand (5):
  - MedLab, Timaru, South Canterbury
  - Timaru Hospital, Timaru, South Canterbury
  - Timaru Rheumatology Studies, Timaru, South Canterbury
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Capital Coast District Health Board, Wellington
- Peru (7):
  - Unidad de Investigacion en Medicina Interna y Enfermedades Criticas, Arequipa
  - Oficina administrativa, Arequipa, Arequipa
  - ABK REUMA SRL-Medicentro Biociencias Peru SRL, Lima
  - Clinica Medica Cayetano Heredia, Lima
  - Centro de Investigación para el Estudio de Enfermedades Reumáticas, Lima
  - Instituto de Ginecología y Reproducción & Cirugía Mínimamente Invasiva, Lima
  - Oficina Administrativa, Lima Lima
- Poland (16):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - NZOZ Zdrowie Osteo-Medic s.c., Bialystok
  - Centrum Kliniczno-Badawcze J.Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - NZOZ Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska Lek. med. Barbara Bazela, Elblag
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Centrum Medyczne Pratia Katowice, Katowice
  - Zespol Poradni Specjalistycznych "REUMED" Filia nr 2, Lublin
  - NZOZ Lecznica MAK-MED. S.C., Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM Dr Hab. Med. Pawel Hrycaj, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej ''Nasz Lekarz'', Torun
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - ''Rheuma Medicus'' Zakład Opieki Zdrowotnej, Warsaw
  - Synexus Polska Sp. z o.o. Oddział we Wroclawiu, Wroclaw
- Russia (14):
  - GBUZ Republican hospital n.a. V.A. Baranov, Petrozavodsk, Republic of Karelia
  - LLC Alliance Biomedical Ural group, Izhevsk
  - GAUZ of Kemerovo Region "Regional clinical hospital for war veterans", Kemerovo
  - GMU Kursk Regional Clinical Hospital of the Healthcare Committee of the Kursk Region, Kursk
  - Municipal Clinical Hospital No. 1 Named after N.I. Pirogov, Moscow
  - GBUZ of city of Moscow City clinical hospital n.a. A.K.Eramishantsev of Ministry of Healthcare of, Moscow
  - Orenburg State Medical Academy, Orenburg
  - Regional Clinical Hospital, Orenburg
  - GBOU VPO Ryazan State Medical University Named after Academician I.P. Pavlov, Ryazan
  - GBU of Ryazan region Regional clinical cardiology dispanser, Ryazan
  - Spb GBUZ "Clinical rheumatology hospital # 25" City CDC prevention of osteoporosis, Saint Petersburg
  - GUZ " Regional clinical hospital", Saratov
  - GBUZ VO Regional clinical hospital, Vladimir
  - GBKUZ of Yaroslavl region "City hospital n. a. N.A. Semashko", Yaroslavl
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy,, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Special Hospital for Rheumatic Diseases Novi Sad, Novi Sad
- South Africa (5):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - St. Augustine's Hospital, Durban, KwaZulu-Natal
  - Arthritis Clinical Research Trials, Dr. C.E Spargo and Dr. R.B Bhorat Practice, Cape Town, Western Cape
  - Panorama Medical Centre, Cape Town, Western Cape
- South Korea (5):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
- Spain (5):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Infanta Luisa, Seville
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
- Ukraine (9):
  - Kyivska miska klinichna likarnia #6, Kyiv
  - Lvivskyi oblasnyi klinichnyi diahnostychnyi tsentr,, Lviv
  - Komunalna 4-a miska klinichna likarnia m. Lvova,, Lviv
  - Komunalnyi zaklad okhorony zdorovia "Kharkivska miska klinichna likarnia #8", M. Kharkiv
  - Komunalnyi zaklad Kyivskoi oblasnoi rady "Kyivska oblasna klinichna likarnia",, M. Kyiv,
  - Bahatoprofilnyi medychnyi tsentr (Universytetska klinika #1), Odesa
  - Komunalnyi zaklad Sumskoi oblasnoi rady "Sumska oblasna klinichna, Sumy
  - Vinnytska oblasna klinichna likarnia im. M.I.Pyrohova revmatolohichne viddilennia, Vinnytsia
  - Komunalna ustanova "Zaporizka oblasna klinichna likarnia" Zaporizkoi oblasnoi rady, Zaporizhzhia
- United Kingdom (4):
  - Basingstoke and North Hampshire Hospital, Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Arrowe Park Hospital, Wirral University Teaching Hospitals NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - Royal United Hospital Bath NHS Foundation Trust ,Royal National Hospital for Rheumatic Diseases, Bath, Somerset
  - The Leeds Institute of Rheumatic and Musculoskeletal Medicine, Leeds, WEST Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kay J, Bock AE, Rehman M, Zhang W, Zhang M, Iikuni N, Alvarez DF. Use of multibiomarker disease activity scores in biosimilarity studies for the treatment of patients with rheumatoid arthritis. RMD Open. 2022 Sep;8(2):e002423. doi: 10.1136/rmdopen-2022-002423. PMID 36180101
- [Derived] Fleischmann RM, Bock AE, Zhang W, Godfrey CM, Vranic I, Cronenberger C, Dokoupilova E. Usability Study of PF-06410293, an Adalimumab Biosimilar, by Prefilled Pen: Open-Label, Single-Arm, Sub-Study of a Phase 3 Trial in Patients with Rheumatoid Arthritis. Rheumatol Ther. 2022 Jun;9(3):839-850. doi: 10.1007/s40744-022-00439-8. Epub 2022 Mar 18. PMID 35304684
- [Derived] Fleischmann RM, Alvarez DF, Bock AE, Cronenberger C, Vranic I, Zhang W, Alten R. Long-term efficacy, safety, and immunogenicity of the adalimumab biosimilar, PF-06410293, in patients with rheumatoid arthritis after switching from reference adalimumab (Humira(R)) or continuing biosimilar therapy: week 52-92 data from a randomized, double-blind, phase 3 trial. Arthritis Res Ther. 2021 Sep 25;23(1):248. doi: 10.1186/s13075-021-02626-4. PMID 34563243
- [Derived] Fleischmann RM, Alvarez DF, Bock AE, Cronenberger C, Vranic I, Zhang W, Alten R. Randomised study of PF-06410293, an adalimumab (ADL) biosimilar, compared with reference ADL for the treatment of active rheumatoid arthritis: results from weeks 26-52, including a treatment switch from reference ADL to PF-06410293. RMD Open. 2021 Apr;7(2):e001578. doi: 10.1136/rmdopen-2021-001578. PMID 33883254
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Fleischmann RM, Alten R, Pileckyte M, Lobello K, Hua SY, Cronenberger C, Alvarez D, Bock AE, Sewell KL. A comparative clinical study of PF-06410293, a candidate adalimumab biosimilar, and adalimumab reference product (Humira(R)) in the treatment of active rheumatoid arthritis. Arthritis Res Ther. 2018 Aug 15;20(1):178. doi: 10.1186/s13075-018-1676-y. PMID 30111357
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5381002&StudyName=A%20Study%20Of%20PF-06410293%20%28Adalimumab-Pfizer%29%20And%20Adalimumab%20%28Humira%29%20In%20Combination%20With%20Methotrexate%20In%20Subjects%20With%20Active%20Rheumatoid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1231 potential participants were screened after signing an informed consent form, of whom 597 participants were randomized to receive study treatment.
Groups:
- PF-06410293/PF-06410293/PF-06410293; Adalimumab-EU/Adalimumab-EU/PF-06410293: Period 1 (first dose to Week 26 predose assessments): participants were blindly randomized in a 1:1 ratio to receive PF-06410293 (a biosimilar to Humira) or adalimumab-EU (Humira from European Union) 40 mg every 2 weeks by subcutaneous injection. All participants randomized into PF-06410293 arm continued to receive PF-06410293 in Periods 2 and 3. Period 2 (Week 26 dosing to Week 52 predose assessments): participants from adalimumab-EU arm were blindly re-randomized in a 1:1 ratio to remain on adalimumab-EU or transition to PF-06410293. Period 3 (Week 52 dosing to Week 78 end of treatment visit): all the remaining participants on adalimumab-EU were switched to open-label PF-06410293.
- Adalimumab-EU/PF-06410293/PF-06410293: Period 1 (first dose to Week 26 predose assessments): participants were blindly randomized in a 1:1 ratio to receive PF-06410293 (a biosimilar to Humira) or adalimumab-EU (Humira from European Union) 40 mg every 2 weeks by subcutaneous injection. [This reporting group in Period 1 is a placeholder box only (not part of the 1:1 randomization).] All participants randomized into PF-06410293 arm continued to receive PF-06410293 in Periods 2 and 3. Period 2 (Week 26 dosing to Week 52 predose assessments): participants from adalimumab-EU arm were blindly re-randomized in a 1:1 ratio to remain on adalimumab-EU or transition to PF-06410293. Period 3 (Week 52 dosing to Week 78 end of treatment visit): all the remaining participants on adalimumab-EU were switched to open-label PF-06410293.
Period: Period 1: First Dose to Week 26 Pre-dose
Arm/Group | PF-06410293/PF-06410293/PF-06410293 | Adalimumab-EU/Adalimumab-EU/PF-06410293 | Adalimumab-EU/PF-06410293/PF-06410293
Started | 297 | 300 | 0
Received Treatment | 297 | 299 | 0
Completed | 293 | 284 | 0
Not Completed | 4 | 16 | 0
Not completed — Insufficient Clinical response | 0 | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 8 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Period: Period 2: Week 26 to Week 52 Pre-dose
Arm/Group | PF-06410293/PF-06410293/PF-06410293 | Adalimumab-EU/Adalimumab-EU/PF-06410293 | Adalimumab-EU/PF-06410293/PF-06410293
Started | 283 | 135 | 134
Received Treatment | 283 | 135 | 133
Completed | 263 | 122 | 127
Not Completed | 20 | 13 | 7
Not completed — Insufficient clinical response | 4 | 1 | 3
Not completed — Non-compliance with study treatment | 0 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 1
Not completed — Adverse Event | 6 | 7 | 3
Not completed — Other | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Period 3: Week 52 Dosing to Week 78
Arm/Group | PF-06410293/PF-06410293/PF-06410293 | Adalimumab-EU/Adalimumab-EU/PF-06410293 | Adalimumab-EU/PF-06410293/PF-06410293
Started | 259 | 121 | 127
Received Treatment | 258 | 120 | 127
Completed | 252 | 118 | 123
Not Completed | 7 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Lost to Follow-up | 4 | 0 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was defined as all participants who were randomized to study treatment.
Groups:
- Period 1: PF-06410293: This reporting group refers to the participants who were randomized to the PF-06410293 group in Period 1, where PF-06410293 40 mg was administered every other week by subcutaneous injection.
- Period 1: Adalimumab-EU: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1, where adalimumab-EU 40 mg was administered every other week by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU | Total
Number analyzed (Participants) | 297 | 300 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.6) | 53.5 (12.9) | 52.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 229 | 470
  Male | 56 | 71 | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 261 | 256 | 517
  Black | 6 | 9 | 15
  Asian | 16 | 17 | 33
  Other | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12: Period 1
Description: ACR20 is a categorical variable indicating a 20% or greater improvement in tender and swollen joint counts and 20% or greater improvement in 3 of the 5 other ACR-core set measures: patient's assessment of arthritis pain (PAAP); patient's global assessment of arthritis (PGA); physician's global assessment of arthritis (PGAA); high sensitivity C-reactive protein (hs-CRP); and Health Assessment Questionnaire - Disability Index (HAQ-DI).
Time Frame: Week 12
Population: The Intent-to-Treat (ITT) population (Period 1) was defined as all participants who were randomized to study treatment. Non-responder imputation was applied.
Measure: Number; unit: percentage of participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
percentage of participants | 68.35 | 71.33
Statistical Analysis 1: Comparison: Period 1: PF-06410293 vs Period 1: Adalimumab-EU; Test type: Non-Inferiority or Equivalence — Confidence interval (CIs) calculated by the score statistic method were used for the inference of the equivalence for ACR20 at Week 12. Therapeutic equivalence could be established if the 2-sided 95% CI fell within (-14%, 14%). Non-responder imputation was applied. Comparisons between treatments were computed as PF-06410293 versus Adalimumab-EU; Week 12 ACR20 response rate difference = -2.98, 95% CI 2-sided [-10.38 to 4.44]
Statistical Analysis 2: Comparison: Period 1: PF-06410293 vs Period 1: Adalimumab-EU; Test type: Non-Inferiority or Equivalence — Confidence interval (CIs) calculated by the score statistic method were used for the inference of the equivalence for ACR20 at Week 12. Therapeutic equivalence could be established if 2-sided 90% CI fell within (-12%, 15%). Non-responder imputation was applied. Comparisons between treatments were computed as PF-06410293 versus Adalimumab-EU; Week 12 ACR20 response rate difference = -2.98, 90% CI 2-sided [-9.25 to 3.28]

2. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Other Time Points Other Than Week 12: Period 1
Description: as for outcome 1
Time Frame: Weeks 2, 4, 6, 8, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: PF-06410293: This reporting group refers to the participants who were randomized to the PF-06410293 group in Period 1. PF-06410293 40 mg was administered every other week by subcutaneous injection in Period 1.
- Period 1: Adalimumab-EU: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1. Adalimumab-EU 40 mg was administered every other week by subcutaneous injection in Period 1.
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Week 2: number analyzed (Participants) | 294 | 295
  Week 2 | 93 | 96
  Week 4: number analyzed (Participants) | 294 | 294
  Week 4 | 154 | 157
  Week 6: number analyzed (Participants) | 295 | 294
  Week 6 | 182 | 179
  Week 8: number analyzed (Participants) | 292 | 293
  Week 8 | 206 | 204
  Week 18: number analyzed (Participants) | 293 | 287
  Week 18 | 232 | 221
  Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Week 26 (pre-dose) | 248 | 234

3. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response: Period 2
Description: as for outcome 1
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Groups:
- Period 2: PF-06410293/PF-06410293: This reporting group refers to the participants who were randomized to the PF-06410293 group in Period 1 and continued to receive PF-06410293 in Period 2. PF-06410293 40 mg was administered every other week by subcutaneous injection in both periods.
- Period 2: Adalimumab-EU/Adalimumab-EU: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1 and remained in the adalimumab-EU group in Period 2. Adalimumab-EU 40 mg was administered every other week by subcutaneous injection in both periods.
- Period 2: Adalimumab-EU/PF-06410293: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1 and switched to PF-06410293 in Period 2. Study drug 40 mg was administered every other week by subcutaneous injection in both periods.
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26: number analyzed (Participants) | 283 | 134 | 134
  Week 26 | 245 | 114 | 116
  Week 30: number analyzed (Participants) | 280 | 132 | 131
  Week 30 | 245 | 111 | 116
  Week 36: number analyzed (Participants) | 275 | 128 | 132
  Week 36 | 236 | 105 | 118
  Week 44: number analyzed (Participants) | 267 | 125 | 130
  Week 44 | 233 | 106 | 108
  Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Week 52 (pre-dose) | 234 | 107 | 113

4. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response: Period 3
Description: as for outcome 1
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Groups:
- Period 3: PF-06410293/PF-06410293/PF-06410293: This reporting group refers to the participants who were randomized to the PF-06410293 group in Period 1 and continued to receive PF-06410293 in Period 2 and Period 3. PF-06410293 40 mg was administered every other week by subcutaneous injection in all 3 periods.
- Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1, remained in the adalimumab-EU group in Period 2 and received PF-06410293 in Period 3. Study drug 40 mg was administered every other week by subcutaneous injection in all 3 periods.
- Period 3: Adalimumab-EU/PF-06410293/PF-06410293: This reporting group refers to the participants who were randomized to the adalimumab-EU group in Period 1 and switched to PF-06410293 from Period 2 and continued on PF-06410293 in Period 3. Study drug 40 mg was administered every other week by subcutaneous injection in all 3 periods.
- Period 3 Total: This reporting group refers to the participants who entered Period 3, where PF-06410293 40 mg was administered every other week by subcutaneous injection.
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Week 52 | 229 | 106 | 112 | 447
  Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Week 56 | 230 | 105 | 106 | 441
  Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Week 66 | 226 | 103 | 108 | 437
  Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Week 76 | 219 | 95 | 106 | 420
  Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Week 78 | 216 | 102 | 109 | 427

5. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) Response: Period 1
Description: ACR50 is a categorical variable indicating a 50% or greater improvement in tender and swollen joint counts and 50% or greater improvement in 3 of the 5 other ACR-core set measures: patient's assessment of arthritis pain (PAAP); patient's global assessment of arthritis (PGA); physician's global assessment of arthritis (PGAA); high sensitivity C-reactive protein (hs-CRP); and Health Assessment Questionnaire - Disability Index (HAQ-DI).
Time Frame: Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Week 2: number analyzed (Participants) | 294 | 295
  Week 2 | 25 | 18
  Week 4: number analyzed (Participants) | 294 | 294
  Week 4 | 53 | 43
  Week 6: number analyzed (Participants) | 295 | 294
  Week 6 | 82 | 82
  Week 8: number analyzed (Participants) | 292 | 293
  Week 8 | 101 | 100
  Week 12: number analyzed (Participants) | 291 | 293
  Week 12 | 118 | 119
  Week 18: number analyzed (Participants) | 293 | 287
  Week 18 | 134 | 141
  Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Week 26 (pre-dose) | 177 | 164

6. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) Response: Period 2
Description: as for outcome 5
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26: number analyzed (Participants) | 283 | 134 | 134
  Week 26 | 175 | 76 | 86
  Week 30: number analyzed (Participants) | 280 | 132 | 131
  Week 30 | 169 | 67 | 82
  Week 36: number analyzed (Participants) | 275 | 128 | 132
  Week 36 | 173 | 70 | 94
  Week 44: number analyzed (Participants) | 267 | 125 | 130
  Week 44 | 182 | 67 | 87
  Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Week 52 (pre-dose) | 178 | 75 | 97

7. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) Response: Period 3
Description: as for outcome 5
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Week 52 | 177 | 74 | 96 | 347
  Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Week 56 | 175 | 78 | 94 | 347
  Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Week 66 | 177 | 75 | 92 | 344
  Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Week 76 | 179 | 66 | 90 | 335
  Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Week 78 | 185 | 71 | 90 | 346

8. Secondary Outcome: Number of Participants With an American College of Rheumatology 70% (ACR70) Response: Period 1
Description: ACR70 is a categorical variable indicating a 70% or greater improvement in tender and swollen joint counts and 70% or greater improvement in 3 of the 5 other ACR-core set measures: patient's assessment of arthritis pain (PAAP); patient's global assessment of arthritis (PGA); physician's global assessment of arthritis (PGAA); high sensitivity C-reactive protein (hs-CRP); and Health Assessment Questionnaire - Disability Index (HAQ-DI).
Time Frame: Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Week 2: number analyzed (Participants) | 294 | 295
  Week 2 | 2 | 6
  Week 4: number analyzed (Participants) | 294 | 294
  Week 4 | 11 | 11
  Week 6: number analyzed (Participants) | 295 | 294
  Week 6 | 24 | 26
  Week 8: number analyzed (Participants) | 292 | 293
  Week 8 | 37 | 35
  Week 12: number analyzed (Participants) | 291 | 293
  Week 12 | 49 | 57
  Week 18: number analyzed (Participants) | 293 | 287
  Week 18 | 64 | 66
  Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Week 26 (pre-dose) | 88 | 93

9. Secondary Outcome: Number of Participants With an American College of Rheumatology 70% (ACR70) Response: Period 2
Description: as for outcome 8
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26: number analyzed (Participants) | 283 | 134 | 134
  Week 26 | 88 | 41 | 52
  Week 30: number analyzed (Participants) | 280 | 132 | 131
  Week 30 | 96 | 41 | 49
  Week 36: number analyzed (Participants) | 275 | 128 | 132
  Week 36 | 102 | 36 | 59
  Week 44: number analyzed (Participants) | 267 | 125 | 130
  Week 44 | 109 | 44 | 53
  Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Week 52 (pre-dose) | 103 | 43 | 59

10. Secondary Outcome: Number of Participants With an American College of Rheumatology 70% (ACR70) Response: Period 3
Description: as for outcome 8
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Week 52 | 103 | 42 | 58 | 203
  Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Week 56 | 101 | 42 | 59 | 202
  Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Week 66 | 112 | 48 | 60 | 220
  Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Week 76 | 118 | 39 | 63 | 220
  Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Week 78 | 128 | 48 | 69 | 245

11. Secondary Outcome: Change From Baseline in Tender Joint Count: Period 1
Description: Sixty-eight (68) joints were assessed by an independent blinded joint assessor to determine the number of joints that were considered tender. The 68 joints assessed were: upper body including temporomandibular, sternoclavicular, acromioclavicular; upper extremity including shoulder, elbow, wrist (radiocarpal, carpal and carpometacarpal considered as 1 unit), metacarpophalangeals (MCP I, II, III, IV, V), thumb interphalangeal, proximal interphalangeals (PIP II, III, IV, V), and distal interphalangeals (DIP II, III, IV, V); lower extremity including hip, knee, ankle, tarsus (subtalar, transverse tarsal and tarsometatarsal considered as 1 unit), metatarsophalangeals (MTP I, II, III, IV, V), great toe interphalangeal, proximal and distal interphalangeals combined (PIP and DIP II, III, IV, V).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
joints
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 24.3 (12.29) | 26.7 (14.80)
  Change at Week 2: number analyzed (Participants) | 294 | 295
  Change at Week 2 | -7.5 (9.89) | -7.1 (9.14)
  Change at Week 4: number analyzed (Participants) | 294 | 294
  Change at Week 4 | -10.2 (10.59) | -10.7 (9.92)
  Change at Week 6: number analyzed (Participants) | 295 | 294
  Change at Week 6 | -12.8 (11.28) | -13.1 (11.93)
  Change at Week 8: number analyzed (Participants) | 292 | 293
  Change at Week 8 | -14.2 (11.37) | -15.2 (11.84)
  Change at Week 12: number analyzed (Participants) | 291 | 293
  Change at Week 12 | -15.4 (11.69) | -16.1 (12.65)
  Change at Week 18: number analyzed (Participants) | 293 | 287
  Change at Week 18 | -16.8 (11.42) | -17.3 (12.69)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Change at Week 26 (pre-dose) | -18.4 (11.41) | -19.2 (12.52)

12. Secondary Outcome: Change From Baseline in Tender Joint Count: Period 2
Description: as for outcome 11
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
joints
  Baseline | 23.7 (11.87) | 26.8 (14.72) | 25.5 (15.00)
  Change at Week 26: number analyzed (Participants) | 283 | 134 | 134
  Change at Week 26 | -18.4 (11.34) | -20.1 (12.47) | -19.3 (11.99)
  Change at Week 30: number analyzed (Participants) | 280 | 132 | 131
  Change at Week 30 | -19.0 (11.85) | -19.5 (14.28) | -19.4 (12.22)
  Change at Week 36: number analyzed (Participants) | 275 | 128 | 132
  Change at Week 36 | -18.7 (12.01) | -20.1 (12.62) | -20.4 (12.56)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -19.4 (12.01) | -21.5 (13.56) | -20.2 (12.94)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Change at Week 52 (pre-dose) | -18.9 (11.49) | -21.0 (14.14) | -21.2 (12.95)

13. Secondary Outcome: Change From Baseline in Tender Joint Count: Period 3
Description: as for outcome 11
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
joints
  Baseline | 23.8 (11.89) | 26.5 (14.97) | 25.4 (14.77) | 24.9 (13.45)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Change at Week 52 | -19.3 (11.38) | -21.2 (14.13) | -21.2 (13.00) | -20.2 (12.50)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -19.4 (11.27) | -21.1 (13.55) | -21.6 (13.43) | -20.4 (12.42)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -19.5 (10.97) | -21.3 (12.83) | -21.6 (13.55) | -20.5 (12.12)
  Change at Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Change at Week 76 | -20.6 (11.75) | -22.0 (14.06) | -22.0 (14.00) | -21.3 (12.89)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -20.5 (11.53) | -21.1 (13.23) | -22.1 (14.26) | -21.1 (12.67)

14. Secondary Outcome: Change From Baseline in Swollen Joint Count: Period 1
Description: Sixty-six (66) joints were assessed for swelling, the same as those listed for tender joint count, excluding the right and left hip joints.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
joints
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 15.4 (7.81) | 17.0 (9.86)
  Change at Week 2: number analyzed (Participants) | 294 | 295
  Change at Week 2 | -5.7 (6.31) | -6.1 (7.23)
  Change at Week 4: number analyzed (Participants) | 294 | 294
  Change at Week 4 | -7.7 (7.04) | -8.2 (8.38)
  Change at Week 6: number analyzed (Participants) | 295 | 294
  Change at Week 6 | -9.0 (7.37) | -9.7 (8.97)
  Change at Week 8: number analyzed (Participants) | 292 | 293
  Change at Week 8 | -9.8 (7.06) | -11.0 (8.50)
  Change at Week 12: number analyzed (Participants) | 291 | 293
  Change at Week 12 | -10.4 (7.38) | -11.8 (8.87)
  Change at Week 18: number analyzed (Participants) | 293 | 287
  Change at Week 18 | -11.3 (6.76) | -13.0 (9.45)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Change at Week 26 (pre-dose) | -12.2 (7.18) | -13.6 (9.12)

15. Secondary Outcome: Change From Baseline in Swollen Joint Count: Period 2
Description: as for outcome 14
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
joints
  Baseline | 15.1 (7.66) | 17.1 (9.60) | 17.0 (10.31)
  Change at Week 26: number analyzed (Participants) | 283 | 134 | 134
  Change at Week 26 | -12.2 (7.11) | -13.6 (8.15) | -14.3 (9.84)
  Change at Week 30: number analyzed (Participants) | 280 | 132 | 131
  Change at Week 30 | -12.3 (7.58) | -13.3 (9.31) | -14.3 (9.70)
  Change at Week 36: number analyzed (Participants) | 275 | 128 | 132
  Change at Week 36 | -12.4 (7.76) | -14.2 (8.74) | -14.6 (9.69)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -12.8 (7.12) | -14.7 (8.87) | -14.8 (9.97)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Change at Week 52 (pre-dose) | -12.6 (6.92) | -14.2 (8.29) | -15.2 (9.82)

16. Secondary Outcome: Change From Baseline in Swollen Joint Count: Period 3
Description: as for outcome 14
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
joints
  Baseline | 15.0 (7.59) | 17.3 (9.77) | 16.8 (10.07) | 16.0 (8.85)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Change at Week 52 | -12.8 (6.87) | -14.4 (8.22) | -15.2 (9.75) | -13.7 (8.05)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -12.9 (6.61) | -14.5 (8.65) | -14.9 (9.65) | -13.8 (8.00)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -13.0 (7.09) | -14.9 (8.37) | -15.2 (9.92) | -14.0 (8.23)
  Change at Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Change at Week 76 | -13.3 (7.12) | -14.9 (8.86) | -15.1 (10.27) | -14.1 (8.44)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -13.4 (7.25) | -15.0 (9.35) | -15.1 (10.24) | -14.2 (8.63)

17. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis (PGAA): Period 1
Description: The investigator assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease symptoms, functional capacity and physical examination, and independent of the participant's reported assessments of PGA (patient's global assessment of arthritis) and PAAP (patient's assessment of arthritis pain). The investigator's response was recorded using a 100 mm visual analog scale (VAS), with the 0 mm end labeled "None" and the 100 mm end labeled "Extreme".
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
units on a scale
  Baseline: number analyzed (Participants) | 296 | 298
  Baseline | 65.0 (15.22) | 66.7 (15.80)
  Change at Week 2: number analyzed (Participants) | 293 | 296
  Change at Week 2 | -20.7 (18.62) | -20.5 (18.87)
  Change at Week 4: number analyzed (Participants) | 293 | 294
  Change at Week 4 | -28.9 (20.24) | -29.0 (18.29)
  Change at Week 6: number analyzed (Participants) | 294 | 294
  Change at Week 6 | -32.6 (21.72) | -33.0 (19.87)
  Change at Week 8: number analyzed (Participants) | 291 | 293
  Change at Week 8 | -35.6 (20.86) | -37.1 (18.97)
  Change at Week 12: number analyzed (Participants) | 291 | 293
  Change at Week 12 | -40.4 (19.01) | -40.5 (19.45)
  Change at Week 18: number analyzed (Participants) | 292 | 287
  Change at Week 18 | -44.2 (18.96) | -44.2 (19.64)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 287 | 278
  Change at Week 26 (pre-dose) | -47.2 (18.68) | -46.5 (19.96)

18. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis (PGAA): Period 2
Description: as for outcome 17
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
units on a scale
  Baseline: number analyzed (Participants) | 282 | 135 | 134
  Baseline | 64.9 (15.21) | 66.3 (15.34) | 67.0 (15.56)
  Change at Week 26: number analyzed (Participants) | 282 | 134 | 134
  Change at Week 26 | -47.7 (18.09) | -45.5 (19.80) | -49.2 (18.77)
  Change at Week 30: number analyzed (Participants) | 280 | 131 | 131
  Change at Week 30 | -47.9 (20.02) | -46.5 (19.52) | -49.6 (18.53)
  Change at Week 36: number analyzed (Participants) | 275 | 129 | 132
  Change at Week 36 | -47.3 (20.22) | -45.4 (19.46) | -49.5 (20.47)
  Change at Week 44: number analyzed (Participants) | 266 | 125 | 130
  Change at Week 44 | -49.1 (18.34) | -46.9 (20.16) | -50.5 (20.50)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 267 | 122 | 129
  Change at Week 52 (pre-dose) | -47.9 (18.89) | -48.4 (17.75) | -52.1 (20.01)

19. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis (PGAA): Period 3
Description: as for outcome 17
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
units on a scale
  Baseline: number analyzed (Participants) | 258 | 121 | 127 | 506
  Baseline | 65.4 (14.57) | 66.4 (15.55) | 67.0 (15.73) | 66.1 (15.09)
  Change at Week 52: number analyzed (Participants) | 257 | 120 | 127 | 504
  Change at Week 52 | -48.9 (17.82) | -48.5 (17.87) | -52.2 (19.62) | -49.7 (18.33)
  Change at Week 56: number analyzed (Participants) | 254 | 121 | 124 | 499
  Change at Week 56 | -50.5 (16.95) | -47.7 (20.00) | -51.6 (21.18) | -50.1 (18.85)
  Change at Week 66: number analyzed (Participants) | 251 | 116 | 122 | 489
  Change at Week 66 | -49.4 (18.93) | -49.1 (18.21) | -51.1 (20.29) | -49.8 (19.09)
  Change at Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Change at Week 76 | -50.9 (17.87) | -49.7 (21.07) | -52.3 (20.57) | -51.0 (19.33)
  Change at Week 78: number analyzed (Participants) | 238 | 113 | 120 | 471
  Change at Week 78 | -52.3 (17.40) | -50.8 (19.42) | -52.5 (19.96) | -52.0 (18.55)

20. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP): Period 1
Description: Participants assessed the severity of their arthritis pain using a 100 mm Visual Analog Scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
units on a scale
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 63.7 (18.42) | 65.9 (19.61)
  Change at Week 2: number analyzed (Participants) | 294 | 296
  Change at Week 2 | -13.1 (18.59) | -13.9 (18.72)
  Change at Week 4: number analyzed (Participants) | 294 | 294
  Change at Week 4 | -18.5 (20.35) | -17.4 (20.30)
  Change at Week 6: number analyzed (Participants) | 295 | 294
  Change at Week 6 | -21.9 (21.92) | -21.7 (22.49)
  Change at Week 8: number analyzed (Participants) | 293 | 293
  Change at Week 8 | -24.8 (24.06) | -25.5 (23.18)
  Change at Week 12: number analyzed (Participants) | 292 | 293
  Change at Week 12 | -28.8 (24.80) | -28.5 (23.91)
  Change at Week 18: number analyzed (Participants) | 293 | 287
  Change at Week 18 | -31.5 (23.69) | -31.4 (25.48)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Change at Week 26 (pre-dose) | -35.1 (24.62) | -33.5 (26.09)

21. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP): Period 2
Description: as for outcome 20
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
units on a scale
  Baseline | 63.5 (18.04) | 65.6 (19.91) | 64.4 (19.37)
  Change at Week 26: number analyzed (Participants) | 283 | 134 | 134
  Change at Week 26 | -35.4 (23.87) | -32.4 (25.68) | -36.0 (26.04)
  Change at Week 30: number analyzed (Participants) | 281 | 132 | 131
  Change at Week 30 | -36.3 (24.86) | -34.1 (26.40) | -37.6 (24.47)
  Change at Week 36: number analyzed (Participants) | 276 | 128 | 132
  Change at Week 36 | -35.5 (25.87) | -34.9 (25.74) | -39.4 (24.87)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -38.6 (25.03) | -35.7 (26.16) | -38.3 (28.05)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Change at Week 52 (pre-dose) | -37.4 (25.09) | -36.8 (24.05) | -40.6 (24.16)

22. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP): Period 3
Description: as for outcome 20
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
units on a scale
  Baseline | 63.5 (17.99) | 66.3 (19.98) | 64.5 (19.05) | 64.4 (18.75)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Change at Week 52 | -38.1 (25.06) | -37.3 (23.93) | -40.6 (23.96) | -38.5 (24.50)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -39.1 (23.87) | -37.7 (25.07) | -40.1 (25.62) | -39.0 (24.57)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -39.8 (24.74) | -39.2 (24.76) | -40.7 (26.42) | -39.9 (25.13)
  Change at Week 76: number analyzed (Participants) | 241 | 110 | 116 | 467
  Change at Week 76 | -41.3 (25.60) | -39.3 (25.95) | -42.4 (25.68) | -41.1 (25.67)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -43.7 (25.17) | -41.4 (25.04) | -42.7 (26.09) | -42.9 (25.34)

23. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis (PGA): Period 1
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participant's response was recorded using a 100 mm visual analog scale (VAS), with the 0 mm end labeled "Very Well" and the 100 mm end labeled "Very Poorly".
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
units on a scale
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 64.4 (19.32) | 68.1 (19.49)
  Change at Week 2: number analyzed (Participants) | 294 | 296
  Change at Week 2 | -13.8 (19.03) | -16.3 (18.30)
  Change at Week 4: number analyzed (Participants) | 294 | 294
  Change at Week 4 | -19.7 (20.85) | -21.2 (21.62)
  Change at Week 6: number analyzed (Participants) | 295 | 294
  Change at Week 6 | -22.2 (22.96) | -23.4 (22.69)
  Change at Week 8: number analyzed (Participants) | 293 | 293
  Change at Week 8 | -25.8 (24.01) | -28.4 (23.17)
  Change at Week 12: number analyzed (Participants) | 292 | 293
  Change at Week 12 | -29.3 (24.72) | -31.5 (24.36)
  Change at Week 18: number analyzed (Participants) | 293 | 287
  Change at Week 18 | -32.2 (24.57) | -34.2 (25.94)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Change at Week 26 (pre-dose) | -36.2 (25.16) | -36.3 (26.21)

24. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis (PGA): Period 2
Description: as for outcome 23
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
units on a scale
  Baseline | 64.2 (19.05) | 67.5 (21.02) | 67.8 (17.59)
  Change at Week 26: number analyzed (Participants) | 283 | 134 | 134
  Change at Week 26 | -36.3 (24.47) | -35.3 (26.02) | -38.8 (25.71)
  Change at Week 30: number analyzed (Participants) | 281 | 132 | 131
  Change at Week 30 | -36.7 (26.11) | -35.5 (27.02) | -41.2 (22.34)
  Change at Week 36: number analyzed (Participants) | 276 | 128 | 131
  Change at Week 36 | -36.4 (26.51) | -36.0 (26.30) | -43.1 (22.31)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -39.4 (25.01) | -36.7 (25.43) | -40.6 (26.49)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Change at Week 52 (pre-dose) | -37.5 (25.88) | -38.6 (24.97) | -44.0 (22.94)

25. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis (PGA): Period 3
Description: as for outcome 23
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
units on a scale
  Baseline | 64.1 (19.02) | 67.5 (21.04) | 68.1 (17.30) | 65.9 (19.17)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Change at Week 52 | -38.3 (25.54) | -39.0 (24.94) | -43.9 (22.79) | -39.9 (24.80)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -39.7 (24.47) | -39.1 (25.61) | -43.4 (25.16) | -40.5 (24.93)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -40.6 (25.04) | -39.7 (24.43) | -43.3 (26.63) | -41.1 (25.29)
  Change at Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Change at Week 76 | -41.7 (26.94) | -40.5 (26.56) | -45.3 (23.51) | -42.3 (26.05)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -43.8 (26.05) | -42.0 (25.09) | -45.4 (24.61) | -43.8 (25.44)

26. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI): Period 1
Description: HAQ-DI assesses the degree of difficulty a participant had experienced during the past week in 8 domains of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each activity category consisted of 2-3 items. For each question in the questionnaire, the level of difficulty was scored from 0 to 3 with 0 representing "no difficulty", 1 as "some difficulty", 2 as "much difficulty", and 3 as "unable to do". Any activity that required assistance from another individual or required the use of an assistive device would adjust to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of scores divided by the number of domains answered. Total possible score range was 0-3 with 0 representing "no difficulty", 1 as "some difficulty", 2 as "much difficulty", and 3 as "unable to do". Higher score indicate more difficulty in performing daily living activities.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
units on a scale
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 1.519 (0.6009) | 1.673 (0.6378)
  Change at Week 2: number analyzed (Participants) | 294 | 296
  Change at Week 2 | -0.254 (0.4018) | -0.288 (0.4383)
  Change at Week 4: number analyzed (Participants) | 294 | 294
  Change at Week 4 | -0.338 (0.4720) | -0.375 (0.4555)
  Change at Week 6: number analyzed (Participants) | 295 | 294
  Change at Week 6 | -0.426 (0.5114) | -0.454 (0.5350)
  Change at Week 8: number analyzed (Participants) | 293 | 293
  Change at Week 8 | -0.480 (0.5253) | -0.520 (0.5457)
  Change at Week 12: number analyzed (Participants) | 292 | 293
  Change at Week 12 | -0.530 (0.5218) | -0.543 (0.5882)
  Change at Week 18: number analyzed (Participants) | 293 | 287
  Change at Week 18 | -0.583 (0.5704) | -0.630 (0.6344)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Change at Week 26 (pre-dose) | -0.654 (0.6262) | -0.674 (0.6618)

27. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI): Period 2
Description: as for outcome 26
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
units on a scale
  Baseline | 1.514 (0.5920) | 1.639 (0.6677) | 1.666 (0.6271)
  Change at Week 26: number analyzed (Participants) | 283 | 134 | 134
  Change at Week 26 | -0.658 (0.6250) | -0.652 (0.6293) | -0.723 (0.6763)
  Change at Week 30: number analyzed (Participants) | 281 | 132 | 131
  Change at Week 30 | -0.681 (0.6379) | -0.650 (0.6673) | -0.772 (0.7113)
  Change at Week 36: number analyzed (Participants) | 276 | 129 | 132
  Change at Week 36 | -0.711 (0.6585) | -0.662 (0.6610) | -0.811 (0.7048)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -0.726 (0.6605) | -0.690 (0.6414) | -0.834 (0.6956)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 267 | 123 | 129
  Change at Week 52 (pre-dose) | -0.700 (0.6776) | -0.729 (0.6359) | -0.840 (0.6861)

28. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI): Period 3
Description: as for outcome 26
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
units on a scale
  Baseline | 1.528 (0.5941) | 1.632 (0.6711) | 1.684 (0.6164) | 1.592 (0.6212)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Change at Week 52 | -0.719 (0.6809) | -0.737 (0.6379) | -0.836 (0.6877) | -0.752 (0.6731)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -0.735 (0.6733) | -0.754 (0.6149) | -0.801 (0.6549) | -0.756 (0.6543)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -0.731 (0.6656) | -0.731 (0.6493) | -0.828 (0.6872) | -0.755 (0.6672)
  Change at Week 76: number analyzed (Participants) | 242 | 110 | 115 | 467
  Change at Week 76 | -0.751 (0.6725) | -0.789 (0.7225) | -0.867 (0.7066) | -0.788 (0.6931)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -0.781 (0.6571) | -0.800 (0.7240) | -0.881 (0.7194) | -0.811 (0.6894)

29. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP): Period 1
Description: Serum samples were analyzed to determine the level of hs-CRP, which was an acute-phase reactant.
Time Frame: Baseline, Weeks1, 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
mg/L
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 21.3 (22.69) | 22.8 (25.26)
  Change at Week 1: number analyzed (Participants) | 290 | 294
  Change at Week 1 | -12.6 (19.84) | -13.4 (24.83)
  Change at Week 2: number analyzed (Participants) | 289 | 291
  Change at Week 2 | -11.5 (19.10) | -13.1 (20.74)
  Change at Week 4: number analyzed (Participants) | 292 | 292
  Change at Week 4 | -11.2 (19.94) | -12.6 (23.16)
  Change at Week 6: number analyzed (Participants) | 295 | 293
  Change at Week 6 | -11.3 (18.73) | -12.6 (24.74)
  Change at Week 8: number analyzed (Participants) | 292 | 292
  Change at Week 8 | -9.1 (22.65) | -12.0 (25.68)
  Change at Week 12: number analyzed (Participants) | 291 | 293
  Change at Week 12 | -9.5 (22.81) | -12.2 (25.59)
  Change at Week 18: number analyzed (Participants) | 292 | 286
  Change at Week 18 | -11.4 (20.67) | -12.3 (26.93)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 288 | 276
  Change at Week 26 (pre-dose) | -11.1 (21.92) | -13.6 (26.47)

30. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP): Period 2
Description: Serum samples were analyzed to determine the level of hs-CRP, which was an acute-phase reactant.
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
mg/L
  Baseline | 21.2 (22.47) | 22.0 (24.51) | 22.3 (25.93)
  Change at Week 26: number analyzed (Participants) | 283 | 133 | 134
  Change at Week 26 | -11.3 (21.70) | -11.2 (27.76) | -15.8 (25.10)
  Change at Week 30: number analyzed (Participants) | 279 | 130 | 131
  Change at Week 30 | -11.3 (19.76) | -10.4 (26.85) | -15.0 (24.50)
  Change at Week 36: number analyzed (Participants) | 276 | 128 | 131
  Change at Week 36 | -10.6 (22.58) | -11.8 (25.41) | -12.5 (30.36)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -9.9 (22.08) | -11.1 (27.01) | -14.8 (26.80)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 267 | 123 | 127
  Change at Week 52 (pre-dose) | -10.6 (20.84) | -11.8 (23.85) | -12.8 (28.49)

31. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP): Period 3
Description: Serum samples were analyzed to determine the level of hs-CRP, which was an acute-phase reactant.
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
mg/L
  Baseline | 20.4 (20.43) | 22.3 (25.30) | 22.7 (26.49) | 21.4 (23.25)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 126 | 505
  Change at Week 52 | -10.7 (20.81) | -11.9 (24.04) | -12.9 (28.57) | -11.5 (23.70)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 125 | 501
  Change at Week 56 | -9.9 (25.29) | -11.7 (26.66) | -14.3 (26.64) | -11.4 (25.97)
  Change at Week 66: number analyzed (Participants) | 255 | 116 | 122 | 493
  Change at Week 66 | -11.1 (21.24) | -9.1 (25.83) | -13.2 (26.97) | -11.2 (23.87)
  Change at Week 76: number analyzed (Participants) | 241 | 109 | 113 | 463
  Change at Week 76 | -12.1 (20.58) | -9.8 (22.03) | -11.9 (28.83) | -11.5 (23.15)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -9.7 (24.68) | -11.9 (22.90) | -13.3 (27.06) | -11.1 (24.90)

32. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (4 Components Based on High-Sensitivity C-Reactive Protein) (DAS28-4 [CRP]): Period 1
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, high-sensitivity C-reactive protein (hs-CRP) and patient's global assessment of arthritis (PGA). DAS28-4 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1) + 0.014 (PGA [mm]) + 0.96. Higher score indicate more disease activity. The possible lowest score is 0.96. The possible highest score is difficult to be determined, due to indeterminable nature of hs-CRP level; assuming hs-CRP level is 0 to 500 mg/L, the possible highest score would be 6.8 (when hs-CRP is 0) to 9.04 (when hs-CRP is 500 mg/L).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
units on a scale
  Baseline: number analyzed (Participants) | 297 | 298
  Baseline | 5.9 (0.87) | 6.1 (0.90)
  Change at Week 2: number analyzed (Participants) | 289 | 289
  Change at Week 2 | -1.2 (0.91) | -1.1 (0.92)
  Change at Week 4: number analyzed (Participants) | 292 | 291
  Change at Week 4 | -1.5 (1.00) | -1.6 (1.01)
  Change at Week 6: number analyzed (Participants) | 295 | 293
  Change at Week 6 | -1.9 (1.19) | -1.9 (1.22)
  Change at Week 8: number analyzed (Participants) | 291 | 292
  Change at Week 8 | -2.0 (1.19) | -2.2 (1.22)
  Change at Week 12: number analyzed (Participants) | 290 | 293
  Change at Week 12 | -2.2 (1.20) | -2.3 (1.26)
  Change at Week 18: number analyzed (Participants) | 292 | 286
  Change at Week 18 | -2.5 (1.20) | -2.6 (1.33)
  Change at Week 26 (pre-dose): number analyzed (Participants) | 288 | 276
  Change at Week 26 (pre-dose) | -2.7 (1.18) | -2.8 (1.31)

33. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (4 Components Based on High-Sensitivity C-Reactive Protein) (DAS28-4 [CRP]): Period 2
Description: as for outcome 32
Time Frame: Baseline, Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
units on a scale
  Baseline | 5.9 (0.85) | 6.1 (0.85) | 6.0 (0.98)
  Change at Week 26: number analyzed (Participants) | 283 | 133 | 134
  Change at Week 26 | -2.7 (1.16) | -2.7 (1.28) | -3.0 (1.25)
  Change at Week 30: number analyzed (Participants) | 279 | 130 | 131
  Change at Week 30 | -2.8 (1.25) | -2.7 (1.31) | -3.1 (1.17)
  Change at Week 36: number analyzed (Participants) | 274 | 126 | 130
  Change at Week 36 | -2.8 (1.29) | -2.8 (1.32) | -3.1 (1.20)
  Change at Week 44: number analyzed (Participants) | 267 | 125 | 130
  Change at Week 44 | -3.0 (1.14) | -2.9 (1.26) | -3.2 (1.21)
  Change at Week 52 (pre-dose): number analyzed (Participants) | 267 | 123 | 127
  Change at Week 52 (pre-dose) | -2.9 (1.23) | -2.9 (1.33) | -3.3 (1.26)

34. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (4 Components Based on High-Sensitivity C-Reactive Protein) (DAS28-4 [CRP]): Period 3
Description: as for outcome 32
Time Frame: Baseline, Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
units on a scale
  Baseline | 5.9 (0.86) | 6.1 (0.86) | 6.0 (0.96) | 6.0 (0.89)
  Change at Week 52: number analyzed (Participants) | 258 | 121 | 126 | 505
  Change at Week 52 | -2.9 (1.21) | -2.9 (1.32) | -3.3 (1.25) | -3.0 (1.26)
  Change at Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Change at Week 56 | -3.0 (1.22) | -2.9 (1.34) | -3.3 (1.29) | -3.0 (1.27)
  Change at Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Change at Week 66 | -3.0 (1.19) | -3.0 (1.34) | -3.3 (1.26) | -3.1 (1.24)
  Change at Week 76: number analyzed (Participants) | 241 | 109 | 113 | 463
  Change at Week 76 | -3.1 (1.18) | -3.0 (1.34) | -3.4 (1.29) | -3.2 (1.25)
  Change at Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Change at Week 78 | -3.2 (1.21) | -3.1 (1.37) | -3.4 (1.39) | -3.2 (1.30)

35. Secondary Outcome: Number of Participants Achieving European League Against Rheumatism (EULAR) Response: Period 1
Description: EULAR response was based on DAS28 EULAR response criteria. Good response was achieved if DAS28 improvement from baseline >1.2 and DAS28 =<3.2. Moderate response was achieved if DAS28 improvement from baseline >0.6 to =<1.2 and DAS28 =<5.1; or DAS improvement from baseline >1.2 and DAS28 >3.2. No response was achieved if DAS improvement from baseline =<0.6 (no matter present DAS28 score); or DAS improvement from baseline >0.6 to =<1.2 and DAS28 >5.1.
Time Frame: Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Week 2: number analyzed (Participants) | 289 | 289
  Week 2: Good response | 18 | 20
  Week 2: Moderate response | 161 | 136
  Week 2: No response | 110 | 133
  Week 4: number analyzed (Participants) | 292 | 291
  Week 4: Good response | 48 | 42
  Week 4: Moderate response | 173 | 168
  Week 4: No response | 71 | 81
  Week 6: number analyzed (Participants) | 295 | 293
  Week 6: Good response | 69 | 65
  Week 6: Moderate response | 178 | 173
  Week 6: No response | 48 | 55
  Week 8: number analyzed (Participants) | 291 | 292
  Week 8: Good response | 93 | 89
  Week 8: Moderate response | 160 | 160
  Week 8: No response | 38 | 43
  Week 12: number analyzed (Participants) | 290 | 293
  Week 12: Good response | 104 | 107
  Week 12: Moderate response | 149 | 149
  Week 12: No response | 37 | 37
  Week 18: number analyzed (Participants) | 292 | 286
  Week 18: Good response | 137 | 132
  Week 18: Moderate response | 134 | 125
  Week 18: No response | 21 | 29
  Week 26 (pre-dose): number analyzed (Participants) | 288 | 276
  Week 26 (pre-dose): Good response | 162 | 147
  Week 26 (pre-dose): Moderate response | 110 | 102
  Week 26 (pre-dose): No response | 16 | 27

36. Secondary Outcome: Number of Participants Achieving European League Against Rheumatism (EULAR) Response: Period 2
Description: as for outcome 35
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26: number analyzed (Participants) | 283 | 133 | 134
  Week 26: Good response | 161 | 67 | 80
  Week 26: Moderate response | 109 | 53 | 45
  Week 26: No response | 13 | 13 | 9
  Week 30: number analyzed (Participants) | 279 | 130 | 131
  Week 30: Good response | 160 | 64 | 83
  Week 30: Moderate response | 106 | 54 | 45
  Week 30: No response | 13 | 12 | 3
  Week 36: number analyzed (Participants) | 274 | 126 | 130
  Week 36: Good response | 158 | 59 | 86
  Week 36: Moderate response | 97 | 60 | 39
  Week 36: No response | 19 | 7 | 5
  Week 44: number analyzed (Participants) | 267 | 125 | 130
  Week 44: Good response | 170 | 62 | 83
  Week 44: Moderate response | 92 | 60 | 45
  Week 44: No response | 5 | 3 | 2
  Week 52 (pre-dose): number analyzed (Participants) | 267 | 123 | 127
  Week 52 (pre-dose): Good response | 169 | 61 | 85
  Week 52 (pre-dose): Moderate response | 86 | 54 | 40
  Week 52 (pre-dose): No response | 12 | 8 | 2

37. Secondary Outcome: Number of Participants Achieving European League Against Rheumatism (EULAR) Response: Period 3
Description: as for outcome 35
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52: number analyzed (Participants) | 258 | 121 | 126 | 505
  Week 52: Good response | 169 | 60 | 85 | 314
  Week 52: Moderate response | 80 | 53 | 39 | 172
  Week 52: No response | 9 | 8 | 2 | 19
  Week 56: number analyzed (Participants) | 255 | 121 | 124 | 500
  Week 56: Good response | 171 | 63 | 84 | 318
  Week 56: Moderate response | 72 | 50 | 36 | 158
  Week 56: No response | 12 | 8 | 4 | 24
  Week 66: number analyzed (Participants) | 253 | 116 | 122 | 491
  Week 66: Good response | 174 | 62 | 86 | 322
  Week 66: Moderate response | 69 | 48 | 33 | 150
  Week 66: No response | 10 | 6 | 3 | 19
  Week 76: number analyzed (Participants) | 241 | 109 | 113 | 463
  Week 76: Good response | 170 | 59 | 81 | 310
  Week 76: Moderate response | 64 | 45 | 27 | 136
  Week 76: No response | 7 | 5 | 5 | 17
  Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Week 78: Good response | 167 | 67 | 89 | 323
  Week 78: Moderate response | 65 | 40 | 26 | 131
  Week 78: No response | 7 | 6 | 5 | 18

38. Secondary Outcome: Number of Participants Achieving Disease Activity Score Remission (DAS <2.6): Period 1
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to each component. The components of the DAS28-4 (CRP) assessment included: tender joint count with 28 joints assessed, swollen joint count with 28 joints assessed, high-sensitivity C-reactive protein (hs-CRP) and patient's global assessment of arthritis (PGA). DAS28-4 (CRP) was calculated as 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 ln(CRP [mg/L] +1) + 0.014 (PGA [mm]) + 0.96. The possible lowest score is 0.96. The possible highest score is difficult to be determined, due to indeterminable nature of hs-CRP level; assuming hs-CRP level is 0 to 500 mg/L, the possible highest score would be 6.8 (when hs-CRP is 0) to 9.04 (when hs-CRP is 500 mg/L). Higher score indicate more disease activity; DAS28-4 (CRP) <2.6 indicates remission.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Baseline | 0 | 0
  Week 2: number analyzed (Participants) | 294 | 297
  Week 2 | 9 | 8
  Week 4: number analyzed (Participants) | 294 | 295
  Week 4 | 20 | 17
  Week 6: number analyzed (Participants) | 295 | 294
  Week 6 | 35 | 34
  Week 8: number analyzed (Participants) | 293 | 293
  Week 8 | 49 | 48
  Week 12: number analyzed (Participants) | 292 | 293
  Week 12 | 63 | 62
  Week 18: number analyzed (Participants) | 293 | 287
  Week 18 | 71 | 81
  Week 26 (pre-dose): number analyzed (Participants) | 289 | 278
  Week 26 (pre-dose) | 87 | 99

39. Secondary Outcome: Number of Participants Achieving Disease Activity Score Remission (DAS <2.6): Period 2
Description: as for outcome 38
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26: number analyzed (Participants) | 283 | 134 | 134
  Week 26 | 86 | 41 | 58
  Week 30: number analyzed (Participants) | 281 | 132 | 131
  Week 30 | 96 | 42 | 51
  Week 36: number analyzed (Participants) | 277 | 129 | 132
  Week 36 | 106 | 41 | 54
  Week 44: number analyzed (Participants) | 267 | 125 | 130
  Week 44 | 109 | 44 | 51
  Week 52 (pre-dose): number analyzed (Participants) | 268 | 123 | 129
  Week 52 (pre-dose) | 107 | 40 | 59

40. Secondary Outcome: Number of Participants Achieving Disease Activity Score Remission (DAS <2.6): Period 3
Description: as for outcome 38
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52: number analyzed (Participants) | 258 | 121 | 127 | 506
  Week 52 | 107 | 39 | 59 | 205
  Week 56: number analyzed (Participants) | 255 | 121 | 125 | 501
  Week 56 | 111 | 46 | 57 | 214
  Week 66: number analyzed (Participants) | 255 | 116 | 122 | 493
  Week 66 | 108 | 52 | 61 | 221
  Week 76: number analyzed (Participants) | 242 | 110 | 116 | 468
  Week 76 | 122 | 45 | 60 | 227
  Week 78: number analyzed (Participants) | 239 | 113 | 120 | 472
  Week 78 | 130 | 51 | 68 | 249

41. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Response：Period 1
Description: Participants were considered to be in ACR/EULAR remission when either of the following criteria was met: scores on the tender joint count, swollen joint count, hs-CRP (mg/dL) and PGA (0-10 cm scale) were all =<1; or the score on the simplified disease activity index (SDAI) was =<3.3. SDAI score was the sum of tender joint count (28), swollen joint count (28), PGA (0-10 cm scale), physician's global assessment of arthritis (PGAA, 0-10 cm scale) and hs-CRP (mg/dL).
Time Frame: Weeks 2, 4, 6, 8, 12, 18 and 26 (pre-dose)
Population: The ITT population (Period 1) was defined as all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 300
Participants
  Week 2 | 2 | 3
  Week 4 | 3 | 5
  Week 6 | 14 | 11
  Week 8 | 16 | 21
  Week 12 | 24 | 24
  Week 18 | 29 | 44
  Week 26 (pre-dose) | 38 | 44

42. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Response: Period 2
Description: as for outcome 41
Time Frame: Weeks 26, 30, 36, 44 and 52 (pre-dose)
Population: The ITT population (Period 2) was defined as all participants who completed the Period 2 randomization call.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 134
Participants
  Week 26 | 38 | 26 | 19
  Week 30 | 50 | 26 | 27
  Week 36 | 49 | 21 | 27
  Week 44 | 56 | 29 | 34
  Week 52 (pre-dose) | 53 | 28 | 35

43. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Response: Period 3
Description: as for outcome 41
Time Frame: Weeks 52, 56, 66, 76 and 78
Population: The ITT population (Period 3) was defined as all participants enrolled in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 259 | 121 | 127 | 507
Participants
  Week 52 | 53 | 27 | 34 | 114
  Week 56 | 63 | 28 | 30 | 121
  Week 66 | 57 | 31 | 29 | 117
  Week 76 | 69 | 27 | 36 | 132
  Week 78 | 77 | 34 | 43 | 154

44. Secondary Outcome: Serum Concentration Versus Time Summary: Period 1
Time Frame: Pre-dose on Days 1, 15, 43, 85 and 183, and at any time during Day 8 visit
Population: The analysis population included all participants who received study drug and provided at least 1 post-dose drug concentration measurement in Period 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 299
ng/mL
  Day 1 (Week 0): number analyzed (Participants) | 295 | 295
  Day 1 (Week 0) | 104.8 (1125.1) | 187.3 (1372.7)
  Day 8 (Week 1): number analyzed (Participants) | 288 | 294
  Day 8 (Week 1) | 3756 (1829.8) | 3488 (1938.2)
  Day 15 (Week 2): number analyzed (Participants) | 293 | 296
  Day 15 (Week 2) | 3349 (1601.0) | 3025 (1729.7)
  Day 43 (Week 6): number analyzed (Participants) | 293 | 292
  Day 43 (Week 6) | 6205 (3525.6) | 5526 (3249.2)
  Day 85 (Week 12): number analyzed (Participants) | 292 | 286
  Day 85 (Week 12) | 7575 (4725.1) | 6531 (4302.5)
  Day 183 (Week 26): number analyzed (Participants) | 286 | 271
  Day 183 (Week 26) | 8244 (5494.6) | 7190 (5402.6)

45. Secondary Outcome: Serum Concentration Versus Time Summary: Period 2
Time Frame: Pre-dose on Days 183, 211, 253 and 365
Population: The analysis population included all participants who received study drug and provided at least 1 post-dose drug concentration measurement in Period 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 133
ng/mL
  Day 183 (Week 26): number analyzed (Participants) | 281 | 133 | 130
  Day 183 (Week 26) | 8346 (5463.5) | 7058 (5174.1) | 7557 (5492.8)
  Day 211 (Week 30): number analyzed (Participants) | 276 | 131 | 131
  Day 211 (Week 30) | 8314 (5728.6) | 6831 (5147.2) | 7626 (5335.7)
  Day 253 (Week 36): number analyzed (Participants) | 266 | 123 | 128
  Day 253 (Week 36) | 8066 (5297.3) | 7063 (5234.2) | 8198 (5627.9)
  Day 365 (Week 52): number analyzed (Participants) | 259 | 122 | 126
  Day 365 (Week 52) | 7491 (4946.9) | 6252 (5054.5) | 8157 (5648.5)

46. Secondary Outcome: Serum Concentration Versus Time Summary: Period 3
Time Frame: Pre-dose on Days 365, 393, 463, 547 and 575
Population: The analysis population included all participants who received study drug and provided at least 1 post-dose drug concentration measurement in Period 3.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 258 | 120 | 127 | 505
ng/mL
  Day 365 (Week 52): number analyzed (Participants) | 257 | 120 | 126 | 503
  Day 365 (Week 52) | 7539 (4933.6) | 6298 (5063.7) | 8157 (5648.5) | 7398 (5184.6)
  Day 393 (Week 56): number analyzed (Participants) | 253 | 117 | 121 | 491
  Day 393 (Week 56) | 7402 (5190.6) | 6261 (4999.6) | 8345 (5255.0) | 7362 (5202.5)
  Day 463 (Week 66): number analyzed (Participants) | 247 | 114 | 118 | 479
  Day 463 (Week 66) | 7364 (5118.5) | 6482 (4879.4) | 8118 (5507.9) | 7340 (5183.0)
  Day 547 (Week 78): number analyzed (Participants) | 246 | 115 | 123 | 484
  Day 547 (Week 78) | 6728 (5003.2) | 6217 (5118.7) | 7388 (5380.7) | 6774 (5134.7)
  Day 575 (Follow-up): number analyzed (Participants) | 240 | 113 | 116 | 469
  Day 575 (Follow-up) | 3355 (3239.2) | 3069 (3393.2) | 3802 (3781.1) | 3397 (3419.7)

47. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (NAb): Period 1
Description: Serum samples were analyzed for the presence or absence of ADA using a semi-quantitative electrochemiluminescent (ECL) assay, and ADA positive was defined as ADA titer >=1.88. Serum samples tested positive for ADA were further analyzed for the presence or absence of NAb using a semi-quantitative cell-based assay, and NAb positive was defined as NAb titer >=0.70.
Time Frame: Baseline up to Week 26 (pre-dose)
Population: The analysis population included all randomized participants who received at least 1 dose of study drug, and had at least 1 ADA measurement in Period 1, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 298
Participants
  ADA | 132 | 151
  NAb: number analyzed (Participants) | 132 | 151
  NAb | 41 | 42

48. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (NAb): Period 2
Description: as for outcome 47
Time Frame: Week 26 dosing up to Week 52 (pre-dose)
Population: The analysis population included all randomized participants who received at least 1 dose of study treatment in Period 1, and received at least 1 dose of study treatment in Period 2, and had at least 1 ADA measurement in Period 2, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 134 | 133
Participants
  ADA | 134 | 73 | 61
  NAb: number analyzed (Participants) | 134 | 73 | 61
  NAb | 46 | 18 | 16

49. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (NAb): Period 3
Description: as for outcome 47
Time Frame: Week 52 dosing up to follow-up visit (Week 92)
Population: The analysis population included all participants enrolled and treated in Period 3 who had at least 1 ADA measurement in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 258 | 120 | 127 | 505
Participants
  ADA: number analyzed (Participants) | 256 | 120 | 126 | 502
  ADA | 119 | 65 | 59 | 243
  NAb: number analyzed (Participants) | 119 | 65 | 59 | 243
  NAb | 54 | 30 | 21 | 105

50. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs for Period 1 were events between first dose of study drug in Period 1 and up to Week 26 pre-dose assessments that were absent before treatment or that worsened relative to pre-treatment state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug. AEs included both serious and non-serious AEs.
Time Frame: Baseline (Day 1) up to Week 26 (pre-dose)
Population: Safety population (Period 1) was defined as all randomized participants who received at least 1 dose of study treatment, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 299
Participants
  All-causality TEAE | 143 | 143
  All-causality SAE | 12 | 13
  Treatment-related TEAE | 55 | 69
  Treatment-related SAE | 5 | 4

51. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs for Period 2 were events between first dose of study drug in Period 2 and up to Week 52 pre-dose assessments that were absent before treatment or that worsened relative to prior state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug. AEs included both serious and non-serious AEs.
Time Frame: Week 26 dosing up to Week 52 (pre-dose)
Population: Safety population (Period 2) was defined as all randomized participants who received at least 1 dose of study treatment in Period 1, and received at least 1 dost of study treatment in Period 2, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 135 | 133
Participants
  All-causality TEAE | 123 | 60 | 51
  All-causality SAE | 4 | 6 | 3
  Treatment-related TEAE | 32 | 22 | 18
  Treatment-related SAE | 2 | 2 | 0

52. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 3
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs for Period 3 were events between first dose of study drug in Period 3 and up to Week 92 visit that were absent before treatment or that worsened relative to prior state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug. AEs included both serious and non-serious AEs.
Time Frame: Week 52 dosing up to follow-up visit (Week 92)
Population: Safety population (Period 3) was defined as all participants enrolled and treated in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 258 | 120 | 127 | 505
Participants
  All-causality TEAE | 110 | 61 | 47 | 218
  All-causality SAE | 9 | 9 | 3 | 21
  Treatment-related TEAE | 27 | 13 | 17 | 57
  Treatment-related SAE | 0 | 3 | 0 | 3

53. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 1
Description: Laboratory evaluation included hematology, clinical chemistry, and urinalysis. Each parameter was evaluated against commonly used and widely accepted criteria. Number of participants with any laboratory abnormality during Period 1 (without regard to baseline abnormality) is presented.
Time Frame: Baseline (Day 1) up to Week 26 (pre-dose)
Population: The analysis population included all randomized participants who received at least 1 dose of study treatment and had laboratory test in Period 1, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU
Number analyzed (Participants) | 297 | 298
Participants | 181 | 180

54. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 2
Description: Laboratory evaluation included hematology, clinical chemistry, and urinalysis. Each parameter was evaluated against commonly used and widely accepted criteria. Number of participants with any laboratory abnormality during Period 2 (without regard to baseline abnormality) is presented.
Time Frame: Week 26 dosing up to Week 52 (pre-dose)
Population: The analysis population included all randomized participants who received at least 1 dose of study treatment in Period 1, and received at least 1 dost of study treatment in Period 2, and had laboratory test in Period 2, analyzed by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293
Number analyzed (Participants) | 283 | 134 | 133
Participants | 171 | 85 | 73

55. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 3
Description: Laboratory evaluation included hematology, clinical chemistry, and urinalysis. Each parameter was evaluated against commonly used and widely accepted criteria. Number of participants with any laboratory abnormality during Period 3 (without regard to baseline abnormality) is presented.
Time Frame: Week 52 dosing up to follow-up visit (Week 92)
Population: The analysis population included all participants enrolled and treated in Period 3 who had laboratory test in Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 | Period 3 Total
Number analyzed (Participants) | 256 | 120 | 126 | 502
Participants | 176 | 77 | 77 | 330

56. Other Pre Specified Outcome: Percentage of Participants Who Achieved Delivery Success in Sub-study
Description: A sub-study was conducted to determine whether participants or their non-healthcare professional caregivers could safely and effectively administer PF-06410293 with the sponsor's prefilled pen (PFP) device.
Time Frame: Weeks 56, 58, 60, 62, 64, 66
Population: The analysis population included all participants in the sub-study.
Measure: Number; unit: percentage of participants
Groups:
- Sub-study: PF-06410293 PFP: Participants received 6 consecutive bi-weekly PF-06410293 doses over a period of 10 weeks (Week 56 to Week 66) using the PFP device provided by the sponsor. The first, third and sixth injections were administered at the study site under the supervision of the investigator or a designated observer. All other injections (the second, fourth and fifth) were administered at home.
Arm/Group | Sub-study: PF-06410293 PFP
Number analyzed (Participants) | 50
percentage of participants
  Week 56 | 100.0
  Week 58: number analyzed (Participants) | 48
  Week 58 | 100.0
  Week 60 | 100.0
  Week 62: number analyzed (Participants) | 49
  Week 62 | 100.0
  Week 64: number analyzed (Participants) | 48
  Week 64 | 100.0
  Week 66: number analyzed (Participants) | 49
  Week 66 | 100.0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to Week 92
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event. MedDRAVersion 20.0 was used for Periods 1 and 2; and Version 20.1 was used for Period 3. AEs were analyzed separately for each period.
Arm/Group | Period 1: PF-06410293 | Period 1: Adalimumab-EU | Period 2: PF-06410293/PF-06410293 | Period 2: Adalimumab-EU/Adalimumab-EU | Period 2: Adalimumab-EU/PF-06410293 | Period 3: PF-06410293/PF-06410293/PF-06410293 | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 | Period 3: Adalimumab-EU/PF-06410293/PF-06410293
All-Cause Mortality (participants affected / at risk) | 0/297 | 1/299 | 0/283 | 0/135 | 0/133 | 0/258 | 1/120 | 0/127
Serious Adverse Events (participants affected / at risk) | 12/297 | 13/299 | 4/283 | 6/135 | 3/133 | 9/258 | 9/120 | 3/127
Other Adverse Events (participants affected / at risk) | 21/297 | 18/299 | 15/283 | 5/135 | 6/133 | 24/258 | 14/120 | 15/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: PF-06410293 (N=297) | Period 1: Adalimumab-EU (N=299) | Period 2: PF-06410293/PF-06410293 (N=283) | Period 2: Adalimumab-EU/Adalimumab-EU (N=135) | Period 2: Adalimumab-EU/PF-06410293 (N=133) | Period 3: PF-06410293/PF-06410293/PF-06410293 (N=258) | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 (N=120) | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 (N=127)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: PF-06410293 (N=297) | Period 1: Adalimumab-EU (N=299) | Period 2: PF-06410293/PF-06410293 (N=283) | Period 2: Adalimumab-EU/Adalimumab-EU (N=135) | Period 2: Adalimumab-EU/PF-06410293 (N=133) | Period 3: PF-06410293/PF-06410293/PF-06410293 (N=258) | Period 3: Adalimumab-EU/Adalimumab-EU/PF-06410293 (N=120) | Period 3: Adalimumab-EU/PF-06410293/PF-06410293 (N=127)
Viral upper respiratory tract infection (Infections and infestations) | 21 (22) | 18 (18) | 15 (17) | 5 (6) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 13 (16) | 3 (3) | 10 (10)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 4 (4) | 2 (2) | 3 (3) | 12 (14) | 11 (11) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.